CLINICAL TRIAL: NCT05950100
Title: Impact of Virtual Reality on the Postoperative Balance of Adolescents With Idiopathic Scoliosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Collaborators: Irmandade Santa Casa de Misericórdia de Porto Alegre (Other)
Responsible Party: Principal Investigator, Francisco Scornavacca, Assistant teacher of the Pediatrics Department, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5.930.492
Record Dates: First submitted 2023-07-05; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Scoliosis Idiopathic
Keywords: Virtual Reality; Postural Balance; Scoliosis; Pediatrics; Postoperative Period; Rehabilitation; Physical Therapy Modalities
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Intervention Model Description: Participants who meet the inclusion criteria will be randomized into 2 groups - virtual reality group (GRV) and control group (GC). Both groups will undergo the same assessments and tests.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: The first researcher who will follow the draw will be blinded to the patients' assessments and to the intervention. The second researcher who will evaluate the two groups will be blind to sampling and intervention. And the immersive virtual reality therapy will be conducted by a third researcher (blinded to sampling and assessments).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants in the control group will not receive the intervention with virtual reality, but they will also receive, on the first postoperative day, the physiotherapeutic care offered by the institution, carried out by the hospital's physiotherapist and with the same duration as the other group (GRV), and constituted by the physiotherapeutic procedures commonly used in the hospital (respiratory physiotherapy maneuvers, kinesiotherapy and walking). During each physiotherapy session, in both groups, the visual analogue scale will be applied.
- Virtual reality group (Experimental): Participants will receive the same care provided by the hospital, in addition to the application of the use of virtual reality
  Interventions: Device: Virtual reality group

INTERVENTIONS:
Device: Virtual reality group — It is composed of the physiotherapeutic procedures usually used in the hospital applied by the institution's physiotherapist, and the immersive virtual reality therapy that will be conducted by a third researcher (blind to the sampling and evaluations). Physiotherapeutic consultations will have the conventional duration offered by the Institution and therapy with virtual reality will last 10 minutes, using the game "Aviãozinho". Both interventions will have a frequency of 2x a day (morning and afternoon shifts), during the period of 4 days.
  Other Names: GRV
  Arms: Virtual reality group

SUMMARY:
The aim of this randomized clinical trial is to evaluate the impact of immersive virtual reality on the static and dynamic balance and functionality of adolescents with idiopathic scoliosis after spinal correction surgery. Secondarily, the objective was: (1) to analyze whether treatment with immersive virtual reality interferes with the hospitalization time of the studied population in relation to the average expected time; (2) to evaluate the impact of the use of immersive virtual reality in relation to the pain reported by adolescents with idiopathic scoliosis in the postoperative period; (3) to evaluate the impact of the use of immersive virtual reality on the functionality and quality of life of the studied population. Participants who meet the inclusion criteria will be randomized into 2 groups - virtual reality group (GRV) and control group (GC). Both groups will be assessed for pain, static and dynamic balance, length of stay, functionality and quality of life. Patients belonging to the virtual reality group will receive the intervention, which will consist of physiotherapeutic procedures usually used in the hospital applied by the institution's physiotherapist, and therapy with immersive virtual reality. The control group will receive only the physiotherapy offered by the hospital.

DETAILED DESCRIPTION:
Introduction: Scoliosis affects between 2% and 4% of the world's pediatric population, among these, 80% have no known cause and belong to the idiopathic type of the disease. Adolescent idiopathic scoliosis (AIS), affecting individuals aged 10 to 18 years, is the most prevalent in the world. In severe cases, when the Cobb angle is greater than 50 degrees in the thoracic region and with a tendency to progression, the recommended treatment is surgery. With surgically promoted structural corrections, symptoms are often triggered, such as changes in balance. In addition to surgically triggered biomechanical changes, impairment of the somatosensory and vestibular systems and impaired neuromuscular control of the trunk, commonly associated with individuals with AIS, can influence the worsening of balance. Being determinant for the performance of different daily functional activities independently, and for the quality of human life, the rehabilitation of static and dynamic balance should be a priority in patients with adolescent idiopathic scoliosis after surgery. With an innovative technology, immersive virtual reality provides a level of realism and immersion greater than other means of virtual reality, making the user's expectations in relation to reality more congruent, and, therefore, being able to expand their motor evolution. In addition to being able to contribute to improving balance, VR is positively associated with the active engagement of individuals, improved posture and reduced apathy in performing care. Therefore, the objective of the present study is to evaluate the impact of using immersive virtual reality on the static and dynamic balance and functionality of adolescents with idiopathic scoliosis after spinal correction surgery. Justification: With the increasing insertion of virtual reality as a therapeutic tool capable of contributing to the evolution of balance and other motor skills in different populations and due to changes in balance that the surgical procedure for scoliosis correction can cause, the importance of conducting a study to assess whether virtual reality interferes with balance recovery in patients undergoing scoliosis surgery. This study may contribute to the identification of a possible treatment for the patient's functional recovery after AIS surgery. Methods: This study is characterized as a double-blind Randomized Clinical Trial with intentional sampling. Data collection will be carried out at the Santa Casa de Misericórdia Hospital Complex in Porto Alegre - Santo Antônio Children's Hospital. The activities involving the study participants will only start after approval of the project by the Research Ethics Committee of the Federal University of Health Sciences of Porto Alegre (CEP-UFCSPA) and the Irmandade da Santa Casa de Misericórdia de Porto Alegre (CEP /ISCMPA). Individuals of both sexes, aged between 11 and 18 years old, diagnosed with adolescent idiopathic scoliosis (AIS) and in the postoperative period of spine correction surgery will be included in the research. Participants who have: moderate to severe cognitive impairment will be excluded from the analysis; difficulty understanding simple orders; other physical conditions that limit trunk movements, orthostasis and/or cause pain; and medical contraindication. Participants who meet the inclusion criteria will be randomized into 2 groups - virtual reality group (GRV) and control group (GC). Data analysis will be presented through descriptive statistics appropriate to the nature and distribution of each variable. The significance level adopted for the study will be 5% (α = 0.05) and the statistical program for data analysis will be SPSS for Windows, version 25.

ELIGIBILITY:
Inclusion Criteria:

* individuals of both sexes;
* aged between 11 and 18 years;
* diagnosed with adolescent idiopathic scoliosis (AIS) and in the postoperative period of spine correction surgery.

Exclusion Criteria:

* moderate to severe cognitive impairment;
* difficulty understanding simple orders;
* other physical conditions that limit trunk movements, orthostasis and/or cause pain;
* medical contraindication.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-06-17 (Actual); Primary Completion 2023-12-29 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Timed Up and Go Test (TUG) | 1st and 4th postoperative day
  Instrument that assesses dynamic balance and functional mobility. The subject starts sitting in a chair, with the back resting on the backrest and arms relaxed on the thigh. TUG measures, in seconds, the time required for the individual to get up from the chair, walk 3 meters, turn around and return to the chair, performing the 3-meter course again.
Change in Romberg Test | 1st and 4th postoperative day
  Its purpose is to assess static balance. To perform the test, the volunteer remains in orthostasis, barefoot, with feet parallel and together, on the ground, arms extended along the body, with eyes closed, remaining in this position for one minute

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | until the 4th postoperative day
  It consists of a scale graduated from 0 to 10. The patient provides a score for his pain in a global way at the time of evaluation in each consultation, which can vary between the two extremes (0 = no pain and 10 = extreme pain). The higher the score, the worse the pain.
Length of stay | Baseline
  Evaluated through analysis of medical records between groups.
Sociodemographic questionnaire | 1st postoperative day
  Prepared exclusively for the study, authored by the author, consisting of questions related to personal data, family history and clinical information of the patient.
Revised Scoliosis Research Society-22 (SRS-22r) | 1st and 4th postoperative day
  This questionnaire has 22 questions divided into ive domains: function/activity, pain, self-image/appearance, mental health and satisfaction with management. Each domain contains ive questions, except the satisfaction with management domain, which contains two questions. Each item can be scored from 1 (worst possible) to 5 (best possible). The function/activity, pain, self-image and mental health domains have a total score ranging from 5 to 25. The satisfaction with management domain has a total score ranging from 2 to 10.
Oswestry Disability Index 2.0 (ODI) | 1st and 4th postoperative day
  Considered an effective method to measure disability in patients with low back pain, high severity and different causes. It is an ordinal instrument, which includes 10 criteria with six response alternatives for each criterion. The scale consists of 10 questions with six alternatives, whose value ranges from 0 to 5.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital da Criança Santo Antônio, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Background] Pasha S, Baldwin K. Are we simplifying balance evaluation in adolescent idiopathic scoliosis? Clin Biomech (Bristol). 2018 Jan;51:91-98. doi: 10.1016/j.clinbiomech.2017.11.011. Epub 2017 Nov 29. PMID 29277028
- [Background] Silva KCVD, Pimentel BN, Santos Filha VAVD. Quantitative and qualitative assessment of body balance in active elderly women and their relation to health in general. Codas. 2020 Nov 13;32(6):e20180246. doi: 10.1590/2317-1782/20202018246. eCollection 2020. English, Portuguese. PMID 33206770
- [Background] Jha KK, Karunanithi GB, Sahana A, Karthikbabu S. Randomised trial of virtual reality gaming and physiotherapy on balance, gross motor performance and daily functions among children with bilateral spastic cerebral palsy. Somatosens Mot Res. 2021 Jun;38(2):117-126. doi: 10.1080/08990220.2021.1876016. Epub 2021 Mar 3. PMID 33655813
- [Background] Ravi DK, Kumar N, Singhi P. Effectiveness of virtual reality rehabilitation for children and adolescents with cerebral palsy: an updated evidence-based systematic review. Physiotherapy. 2017 Sep;103(3):245-258. doi: 10.1016/j.physio.2016.08.004. Epub 2016 Sep 27. PMID 28109566
- [Background] Beani E, Filogna S, Martini G, Barzacchi V, Ferrari A, Guidi E, Menici V, Cioni G, Sgandurra G. Application of Virtual Reality Rehabilitation System for the assessment of postural control while standing in typical children and peers with neurodevelopmental disorders. Gait Posture. 2022 Feb;92:364-370. doi: 10.1016/j.gaitpost.2021.12.008. Epub 2021 Dec 10. PMID 34923256
- [Background] Cheng JC, Castelein RM, Chu WC, Danielsson AJ, Dobbs MB, Grivas TB, Gurnett CA, Luk KD, Moreau A, Newton PO, Stokes IA, Weinstein SL, Burwell RG. Adolescent idiopathic scoliosis. Nat Rev Dis Primers. 2015 Sep 24;1:15030. doi: 10.1038/nrdp.2015.30. PMID 27188385
- [Background] Negrini S, Donzelli S, Aulisa AG, Czaprowski D, Schreiber S, de Mauroy JC, Diers H, Grivas TB, Knott P, Kotwicki T, Lebel A, Marti C, Maruyama T, O'Brien J, Price N, Parent E, Rigo M, Romano M, Stikeleather L, Wynne J, Zaina F. 2016 SOSORT guidelines: orthopaedic and rehabilitation treatment of idiopathic scoliosis during growth. Scoliosis Spinal Disord. 2018 Jan 10;13:3. doi: 10.1186/s13013-017-0145-8. eCollection 2018. PMID 29435499
- [Background] Akbar M, Almansour H, Lafage R, Diebo BG, Wiedenhofer B, Schwab F, Lafage V, Pepke W. Sagittal alignment of the cervical spine in the setting of adolescent idiopathic scoliosis. J Neurosurg Spine. 2018 Nov 1;29(5):506-514. doi: 10.3171/2018.3.SPINE171263. Epub 2018 Aug 24. PMID 30141764
- [Background] Marinho, M.F.; Paz, J.V.C. da Qualidade de vida após tratamento cirúrgico para escoliose idiopática do adolescente: revisão sistemática da literatura. Research, Society and Development, v. 11, n. 4, p. e21211427014, 2022.
- [Background] Santiago, H.A.R. A influência da escoliose idiopática do adolescente e do seu tratamento cirúrgico sobre o equilíbrio semi- estático. Teses.Usp.Br, v. 126, n. 16, p. 2016, 2011.
- [Background] Latorre, B.P.; Carvalho, M.T.X.; et al. A realidade virtual melhora o equilíbrio e o desempenho motor de uma criança com paralisia cerebral: relato de caso. Saúde (Santa Maria), v. 46, n. 2, p. 1-8, 2020.
- [Background] Aroeira RMC, Leal JS, Pertence AEM, Casas EBL, Greco M. Non-ionizing method of screening adolescent idiopathic scoliosis in schoolchildren. Cien Saude Colet. 2019 Feb;24(2):523-534. doi: 10.1590/1413-81232018242.12882017. English, Portuguese. PMID 30726384
- [Background] Herdea A, Dragomirescu MC, Ulici A, Lungu CN, Charkaoui A. Controlling the Progression of Curvature in Children and Adolescent Idiopathic Scoliosis Following the Administration of Melatonin, Calcium, and Vitamin D. Children (Basel). 2022 May 21;9(5):758. doi: 10.3390/children9050758. PMID 35626935
- [Background] Herdea A, Stancu TA, Ulici A, Lungu CN, Dragomirescu MC, Charkaoui A. Quality of Life Evaluation Using SRS-30 Score for Operated Children and Adolescent Idiopathic Scoliosis. Medicina (Kaunas). 2022 May 18;58(5):674. doi: 10.3390/medicina58050674. PMID 35630090
- [Background] Gur G, Ayhan C, Yakut Y. The effectiveness of core stabilization exercise in adolescent idiopathic scoliosis: A randomized controlled trial. Prosthet Orthot Int. 2017 Jun;41(3):303-310. doi: 10.1177/0309364616664151. Epub 2016 Sep 13. PMID 27625122
- [Background] Xavier, M.J.; Rodrigues, N.M.N.M.; et al. Realidade virtual na reabilitação da paralisia cerebral: Um estudo de caso. Brazilian Journal of Development, v. 6, n. 7, p. 47002-47011, 2020.
- [Background] Souza Filho, B.A.B. de; Tritany, É.F. Realidade virtual imersiva nos Cuidados Paliativos: perspectivas para a Reabilitação Total. Cadernos Brasileiros de Terapia Ocupacional, v. 30, p. 1-13, 2022.
- [Background] Nicolini-Panisson RD, Donadio MV. Timed "Up & Go" test in children and adolescents. Rev Paul Pediatr. 2013 Sep;31(3):377-83. doi: 10.1590/S0103-05822013000300016. PMID 24142322
- [Background] Silva, B.C.; Torre, C.R.M.A. De; et al. Compensações realizadas por crianças com paralisia cerebral espástica durante o levantar da cadeira. Revista Neurociências, v. 29, p. 1-20, 2021.
- [Background] Melo RS, Marinho SEDS, Freire MEA, Souza RA, Damasceno HAM, Raposo MCF. Static and dynamic balance of children and adolescents with sensorineural hearing loss. Einstein (Sao Paulo). 2017 Jul-Sep;15(3):262-268. doi: 10.1590/S1679-45082017AO3976. PMID 29091145
- [Background] Ries LG, Michaelsen SM, Soares PS, Monteiro VC, Allegretti KM. Cross-cultural adaptation and reliability analysis of the Brazilian version of Pediatric Balance Scale (PBS). Rev Bras Fisioter. 2012 Jun;16(3):205-15. doi: 10.1590/s1413-35552012005000026. Epub 2012 Jun 14. English, Portuguese. PMID 22699691
- [Background] Sá, C. dos S.C. de; Fávero, F.M.; et al. Versão brasileira da Segmental Assessment of Trunk Control (SATCo). Fisioterapia e Pesquisa, v. 24, n. 1, p. 89-99, 2017.
- [Background] CRUZ, D.M.C. da; PARKINSON, S.; et al. Correlações entre a Participação Ocupacional, Independência e Cognição em Adultos com Deficiência Física. Revista Brasileira de Educação Especial, v. 27, p. 105-118, 2021.